CLINICAL TRIAL: NCT06459037
Title: Comparison of Salivary Neuropilin-1 (NRP-1), Cotinine and C-Reactive Protein (CRP) Levels With Periodontal Clinical Parameters in Smokers and Non-Smokers With Different Periodontal Diseases
Brief Title: Comparison of Salivary Biormarkers Levels With Periodontal Clinical Parameters in Smokers and Non-Smokers With Different Periodontal Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Izmir Katip Celebi University (Other)
Responsible Party: Principal Investigator, Şeyma Gündoğdu, Research Assistant at Periodontology, Izmir Katip Celebi University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-TDU-DİŞF-0001
Record Dates: First submitted 2024-06-10; First posted 2024-06-14 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Periodontal Diseases
Keywords: periodontitis; gingivitis; neuropilin-1; crp; cotinine; smoking; biomarker; saliva; salivary; ELISA
MeSH Terms: conditions — Periodontal Diseases; Periodontitis; Gingivitis; Smoking

STUDY DESIGN:
Intervention Model Description: According to full-mouth clinical periodontal measurements including probing depth (PD), clinical attachment level (CAL),bleeding on probing (BOP), gingival index (GI) and plaque index (PI) samples of saliva were obtained from 60 systemically healthy non-smoker individuals with periodontitis (P, n=20), gingivitis(G, n=20) and healthy periodontium (S, n=20) and with 20 systemically healthy smoker individuals with periodontitis (PS, n=20).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Healthy Periodontium (Experimental): Individuals with less than 10% bleeding on probing, probing depth less than 4 mm, and no attachment loss, based on evaluation in 6 areas of each tooth.
  Interventions: Diagnostic Test: Saliva obtaining
- Gingivitis (Experimental): Individuals who, in the evaluation made in 6 areas of each tooth, had bleeding on probing in more than 10% of the areas, had a probing depth of less than 4 mm and had no attachment loss.
  Interventions: Diagnostic Test: Saliva obtaining
- non-smoker periodontitis (Experimental): Individuals who have bleeding on probing in 30% or more of the area, who have a probing pocket depth of 5 mm or more in at least 2 non-adjacent teeth in each quadrant of the jaw, who have attachment loss of 4 mm or more, and who have coronal 1/3 or more (horizontal and/or vertical) bone loss on radiographs.
  Interventions: Diagnostic Test: Saliva obtaining
- smoker periodontitis (Experimental): Individuals who smoke at least 10 cigarettes per day, have bleeding on probing in 30% or more of the area, have a probing pocket depth of 5 mm or more in at least 2 non-adjacent teeth in each quadrant of the jaw, have attachment loss of 4 mm or more, and have coronal 1/3 or more (horizontal and/or vertical) bone loss on radiographs.
  Interventions: Diagnostic Test: Saliva obtaining

INTERVENTIONS:
Diagnostic Test: Saliva obtaining — The patient was asked to sit upright and tilt his/her head forward to collect saliva samples. İn this way, unstimulated saliva was allowed to accumulate in the floor of the mouth. The accumulated saliva was collected in a sterile container. It was then transferred to a propylene tube. The tubes were centrifuged and the clear part at the top of the tube was taken with a sterile syringe and transferred to a different propylene tube with 0.5 ml in each tube. Tubes were stored at -80ºC until the day of analysis.

SUMMARY:
To better understand the pathogenesis of chronic inflammatory diseases, the levels of various cytokines are commonly analyzed in tissues and biological fluids collected from the body. The role of the glycoprotein neuropilin-1 (NRP-1) in inflammatory diseases, as well as the relationship between smoking and periodontal diseases, has been investigated in several studies.

The primary aim of this study is to evaluate the salivary levels of NRP-1 in systemically healthy individuals, including non-smokers with periodontal health, non-smokers with gingivitis, non-smokers with periodontitis, and smokers with periodontitis. Additionally, the study aims to compare the concentration of NRP-1 with C-reactive protein (CRP) levels across these groups to assess potential associations.

A secondary objective is to determine the impact of nicotine exposure by measuring salivary cotinine levels and exploring their relationship with the clinical and biochemical parameters assessed. The study will include a total of 80 participants, divided into four equal groups: 20 non-smokers with periodontal health, 20 patients with gingivitis, 20 non-smokers with periodontitis, and 20 smokers with periodontitis.

For all participants, comprehensive oral clinical parameters will be recorded, and unstimulated saliva samples will be collected. The concentrations of NRP-1, cotinine, and CRP in these samples will be determined using enzyme-linked immunosorbent assay (ELISA). Statistical analyses will then be conducted to evaluate differences in biomarker levels among the groups.

Significant variations in these biomarker levels may indicate that NRP-1 has potential utility as a diagnostic biomarker for periodontal diseases or as a marker to guide treatment strategies. Furthermore, the findings may contribute to a deeper understanding of the interplay between periodontitis and smoking.

DETAILED DESCRIPTION:
The aim of this clinical study is to compare the levels of salivary Neuropilin-1 (NRP-1), cotinine, and C-reactive protein (CRP) among smokers and non-smokers who are systemically and periodontally healthy, as well as those with gingivitis and periodontitis, and to correlate these biomarkers with periodontal clinical parameters. The ultimate goal is to determine the potential impact of smoking on periodontal health and disease through these biomarkers.

"Periodontal diseases" encompass a range of chronic inflammatory conditions affecting the gingiva, alveolar bone, and periodontal ligaments. The process begins with gingivitis, characterized by sulcular pathogenic bacterial accumulation in the gingiva, and can progress to periodontitis, involving impaired host immune response and destruction of connective tissue attachment. Inflammation in affected tissues, degradation of connective tissue, and biochemical signaling in alveolar bone remodeling contribute to the observed clinical morbidity.

Plaque-induced gingivitis is a reversible inflammatory condition resulting from microbial biofilm accumulation on teeth and inadequate removal. It is characterized by gingival redness, swelling, and a tendency to bleed easily. With proper oral hygiene measures, it can resolve spontaneously within approximately one week. In susceptible individuals, gingivitis may progress to periodontitis. Periodontitis is characterized by connective tissue attachment loss and alveolar bone destruction following an inflammatory host response to periodontal pathogens. These destructions lead to the formation of pathological pockets, increased mobility, chewing dysfunction, patient discomfort, and ultimately tooth loss.

The role of specific bacterial species clusters in periodontal disease has been studied using various methods, from classical cultural techniques to molecular, genomic, and proteomic approaches. Certain bacterial species, such as Porphyromonas gingivalis, Tannerella forsythensis, and Treponema denticola, are commonly associated with periodontal disease. As periodontal disease progresses, the number of gram-negative and anaerobic bacteria in dental plaque increases. However, the presence of microbial biofilm alone may not be sufficient for disease development. The disease arises when the balance between microbial biofilm and host response is disrupted, leading to dysbiosis or an excessive immune response to microbial presence.

During periodontal infection, the release of bacterial leukotoxins, collagenases, fibrinolysins, and other proteases contributes to tissue destruction. Epithelial cells serve as a physical barrier against pathogens and initiate innate and adaptive immune responses. Dendritic Langerhans cells in the epithelium capture microbial antigens and transport them to lymphoid tissue for presentation to lymphocytes. This is followed by infiltration of neutrophils, granulocytes, and lymphocytes into the periodontal lesion. Neutrophils attempt to phagocytose and eliminate bacteria but may be insufficient against the size and chronic persistence of microbial biofilm. This intense chronic inflammatory response leads to alveolar bone resorption by osteoclasts and degradation of connective tissue fibers by matrix metalloproteinases, resulting in granulation tissue formation.

Neuropilins are transmembrane glycoproteins expressed in all vertebrates, with NRP-1 and NRP-2 identified as two distinct genes. NRP-1 is located on chromosome 10p12, while NRP-2 is on chromosome 2. Both genes contain 17 exons.Neuropilins lack intracellular tyrosine kinase domains but possess a large extracellular region and a short cytoplasmic tail of approximately 40 amino acids. Neuropilins regulate various functions, including homeostasis, angiogenesis, arteriogenesis, immune regulation, inflammation, cell migration during inflammation, communication with immune cells, cancer, and autoimmune diseases. NRP-1 enhances antigen presentation by facilitating interactions between dendritic cells and T cells. It is expressed in macrophages, dendritic cells, and especially T cells. NRP-1 has been shown to play a role in regulating vascular endothelial cell migration. Additionally, NRP-1 is involved in bone homeostasis and is expressed in osteoblasts and osteoclasts. NRP-1 serves as a receptor for Semaphorin-3A (SEMA3A), Vascular Endothelial Growth Factor-A (VEGF-A), VEGF-B, Placenta Growth Factor (PIGF), and microRNAs.

In periodontitis, there is an immune response against periodontal pathogens involving innate and adaptive immunity, which may include NRP-1 in the interaction between dendritic cells and T cells. An imbalance or dysregulation of this immune response leads to excessive tissue damage and irreversible destruction of dental support.

During acute inflammation, various cells, including macrophages, fibroblasts, and endothelial cells, release pro-inflammatory cytokines such as IL-6, TNF-α, IL-1β, and IL-22. These cytokines stimulate the liver to produce acute-phase proteins (APPs), including serum amyloid A (SAA) and C-reactive protein (CRP). CRP levels increase rapidly within 24 to 72 hours in response to inflammation or tissue damage and decrease after resolution of inflammation or infection. Elevated CRP levels have been linked to various inflammatory conditions, including periodontal diseases.

Saliva contains various components, including electrolytes, epithelial cells, antimicrobial peptides, and enzymes. Salivary analysis has shown potential diagnostic properties for identifying periodontal disease biomarkers. Saliva is considered an attractive diagnostic fluid for oral-related diseases due to its non-invasive collection, ease of obtaining, and presence of various biomarkers.

The study involves systemically healthy 80 participants, including 20 non-smoking individuals with healthy periodontium; 20 individuals with gingivitis; 20 individuals with periodontitis; and 20 smoking individuals with periodontitis. Saliva samples were collected from all participants to analyze the levels of NRP-1, cotinine, and CRP using ELISA (enzyme-linked immunosorbent assay) methods. Clinical periodontal parameters such as probing pocket depth (PPD), clinical attachment level (CAL), bleeding on probing (BOP), and plaque index (PI) were also recorded.

Cotinine, the major metabolite of nicotine, is widely used as a biomarker of tobacco exposure due to its longer half-life (approximately 17 hours) compared to nicotine. Cotinine levels in saliva, serum, or urine can reflect both active and passive tobacco exposure, making it a reliable indicator for quantifying smoking status and intensity.

Smoking is a well-established modifiable risk factor for periodontal disease. It has been shown to alter host immune responses to microbial challenges in the oral cavity. Smoking affects various immune cell functions, such as reducing neutrophil and fibroblast activity, impairing immunoglobulin G (IgG) production, and decreasing the release of growth factors. On the other hand, it increases the expression of pro-inflammatory cytokines like PGE2, IL-1β, IL-6, IL-7, IL-8, IL-10, and IL-15, as well as the prevalence of periodontal pathogens.

Nicotine and its metabolites also affect the oral environment by increasing bacterial colonization on epithelial cells and reducing oxidative potential, promoting anaerobic conditions that favor pathogenic bacteria. These changes accelerate the progression of periodontal disease and complicate its management.

Interestingly, clinical signs of inflammation such as bleeding on probing may appear reduced in smokers due to the vasoconstrictive effects of nicotine, which limits gingival blood flow, edema, and visual signs of inflammation. Despite this, the underlying periodontal destruction may be more severe and progress unnoticed.

Although the relationship between salivary CRP levels and periodontal disease has been studied previously, there is a lack of data in the current literature regarding salivary NRP-1 levels in smoking individuals with periodontal disease. This study aims to fill that gap by examining how salivary levels of NRP-1, cotinine, and CRP vary in smokers versus non-smokers across different periodontal health statuses, and by determining whether NRP-1 can serve as a potential biomarker for periodontal disease progression influenced by smoking.

In conclusion, this study seeks to elucidate the diagnostic and prognostic significance of salivary NRP-1, cotinine, and CRP levels, particularly in the context of smoking and its effect on periodontal health. These findings may contribute to improved risk assessment and personalized approaches in periodontal diagnosis and treatment planning.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy (Determination of volunteers will be based on patient statements in the anamnesis. No additional examination will be performed.)
* At least 16 permanent teeth in the mouth
* For non-smoking groups: never smoked
* For the smoking group: smoking at least 10 cigarettes per day
* No continuously used medications
* No use of antibiotics, anti-inflammatory drugs, and systemic corticosteroids in the last 6 months
* Not pregnant or breastfeeding
* No periodontal treatment in the last 6 months
* For the Periodontitis group: based on the evaluation of 6 sites per tooth, ≥30% bleeding on probing, probing depth ≥5 mm and clinical attachment loss ≥4 mm in at least 2 non-adjacent teeth in a quadrant, and radiographic bone loss of coronal 1/3 or more (horizontal and/or vertical)
* For the Gingivitis group: based on the evaluation of 6 sites per tooth, ≥10% bleeding on probing, probing depth <4 mm, and no clinical attachment loss
* For the Healthy group: based on the evaluation of 6 sites per tooth, <10% bleeding on probing, probing depth <4 mm, and no clinical attachment loss

Exclusion Criteria:

* Any oral or systemic disease
* Regularly using a systemic medication
* During pregnancy or lactation
* Received periodontal treatment within the last 6 months.
* Those who received antibiotic, anti-inflammatory or systemic corticosteroid medication in the last 6 months

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2024-05-10 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2025-03-20 (Actual)

PRIMARY OUTCOMES:
salivary CRP level | 24 hours after taking the clinical measurements at the first visit
  The total amount of CRP in saliva
Salivary Neuropilin-1 level | 24 hours after taking the clinical measurements at the first visit
  The total amount of Neuropilin-1(NRP-1) in saliva
Salivary Cotinine level | 24 hours after taking the clinical measurements at the first visit
  The total amount of , Cotinine in saliva

SECONDARY OUTCOMES:
Periodontal Probing Depth | Day 1 (first visit)
  With the help of a periodontal probe, the distance between the gingival margin and the sulcus/pocket base will be measured from six points of the tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal/lingual, mid buccal/palatinal and distobuccal/palatinal. During the measurement, care will be taken to ensure that the probe is parallel to the long axis of the tooth and that excessive force is not applied. The values will be summed and divided by 6 to calculate the average PPD for each patient.
Clinical Attachment Level | Day 1 (first visit)
  With the help of a periodontal probe, the distance between the enamel-cement border and the sulcus/pocket base will be measured at six points of the tooth: mesiobuccal, midbuccal, distobuccal, mesiopalatinal/lingual, mid buccal/palatinal and distobuccal/palatinal. The values will be summed and divided by 6 to calculate the average amount of clinical attachment level for each patient.
Plaque Index | Day 1 (first visit)
  For Silness&Löe plaque index measurement, values will be obtained from four surfaces of each tooth: mesial, distal, vestibular and palatinal. The values will be summed and divided by four to determine the PI score for each tooth. Scoring will be done as follows; 0: No bacterial plaque on the gingival area of the tooth surface. 1: No bacterial plaque is visible on the surface of the tooth by eye, but after probing, bacterial plaque is observed at the tip of the probe. 2: The gingival area is covered with a thin to moderate amount of bacterial plaque, which is visible by eye. 3: There is a large amount of soft debris, the thickness of which completely fills the gingival groove and the interdental space is filled with soft debris.
Bleeding on Probing | Day 1 (first visit)
  The following index criteria will be used to determine the degree of inflammation in the soft tissue surrounding the vestibular, lingual, mesial and distal surfaces of all teeth. The number of positive (+) scoring areas on the examined surfaces will be calculated as a percentage of the total number of examined areas. (-): No bleeding when the periodontal probe is passed along the gingival sulcus. (+): Bleeding is present at the gingival margin.
Gingival Index | Day 1 (first visit)
  According to Löe&Silness gingival index; vestibule, lingual, mesial and distal surfaces of all teeth will be examined. The values will be summed and divided by four to determine the GI score for each tooth. 0: Healthy gingiva. 1: Mild inflammation, mild discoloration and edema but no bleeding after probing. 2: Moderate inflammation, edema, redness and brightness, bleeding on probing. 3: Severe inflammation and redness, edema, ulceration and tendency to spontaneous bleeding.

CONTACTS AND LOCATIONS:
Overall Officials: Abdullah Seçkin Ertuğrul, Prof. Dr., Study Director — Izmir Katip Çelebi University, Faculty of Dentistry, Department of Periodontology
Locations (1):
- Izmir Katip Çelebi University Department of Periodontology, Izmir, Çiğli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No